CLINICAL TRIAL: NCT05153382
Title: Dialectical Behavior Therapy for Youth With and/or at Familial Risk for Bipolar Disorder: Focus on Predictors and Mediators of Treatment Outcomes
Brief Title: Dialectical Behavior Therapy for Youth With and/or at Familial Risk for Bipolar Disorder
Acronym: DB1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Benjamin Goldstein, Director of the Centre for Youth Bipolar Disorder, Clinician-Scientist, Professor of Psychiatry, Pharmacology & Toxicology, and Psychological Clinical Science, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 049/2021
Record Dates: First submitted 2021-11-05; First posted 2021-12-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Bipolar Disorder
Keywords: Youth; Dialectical Behavior Therapy (DBT)
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth with and/or at familial risk for bipolar disorder (Experimental): 60 youth aged 13 to 23 with and/or at familial risk for bipolar disorder will be enrolled in the dialectical behavioral therapy intervention.
  Interventions: Behavioral: Dialectical behavioral therapy

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy — DBT will be conducted over 1 year, and divided into two modalities: skills training, conducted in 60 minute biweekly meetings and individual therapy conducted in 60 minute biweekly sessions. Family participation in skills training is highly encouraged. Skills training proceeds as follows: psychoeducation, mindfulness skills, emotion regulation skills, distress tolerance skills, interpersonal skills, and walking the middle path skills. Individual therapy sessions aim to aid the youth in applying skills in their daily lives. We adopt the standard DBT hierarchy of treatment targets, whereby the individual therapist selects behaviors to focus on based on the following priorities: 1) decreasing life-threatening behaviors, 2) decreasing therapy-interfering behaviors, 3) decreasing quality-of-life interfering behaviors, and 4) increasing behavioral skills. Therapists will be available to participants by cell phone for in-vivo skills coaching between sessions.
  Other Names: DBT

SUMMARY:
Dialectical behavior therapy (DBT) will be conducted over 1 year in youth with and/or at familial risk for bipolar disorder (BD). DBT will be divided into two modalities: 1) DBT skills training; and 2) DBT individual therapy sessions. Skills training sessions will incorporate the 5 standard adolescent DBT modules: mindfulness skills, emotion regulation skills, distress tolerance skills, interpersonal skills, and walking the middle path skills and an additional module on psychoeducation about DBT and BD. This study seeks to build upon the knowledge base in this area by offering DBT to youth with and/or at familial risk for BD with an emphasis on predictors and mediators of treatment outcomes.

DETAILED DESCRIPTION:
In recent years, studies led by investigators at the University of Pittsburgh have emerged that demonstrate the promise of adapting dialectical behavior therapy (DBT) to align with the unique needs of youth with bipolar disorder (BD). Our group has conducted a dissemination and implementation DBT study at Sunnybrook Health Sciences Centre focused specifically on youth with BD. Preliminary data from that study demonstrate that the study therapists, now at CAMH, have achieved fidelity and competence in delivering the intervention, as evidenced by adherence coding scores and participant outcomes. The DBT intervention is based on Miller et al.'s DBT for suicidal adolescents, with modifications for youth with BD. A co-investigator on this study, Dr. T. Goldstein, developed and refined the manualized treatment during her National Institute of Mental Health K23 award in consultation with Dr. Miller. In keeping with the protocol implemented in prior studies, DBT in the present study will be conducted over 1 year, and divided into two modalities: 1) DBT skills training (approximately 60 minute biweekly meetings); and 2) DBT individual therapy sessions (approximately 60 minute biweekly sessions) alternating with skills training. Family involvement in skills training will be strongly encouraged, but not mandatory. Master's level therapists with clinical experience in youth with BD and their families will conduct DBT. This study includes 1 year of assessments (intake, 3, 6, 9, and 12 months) while the intervention is being delivered. The target sample size will be 60 youth with and/or at familial risk for BD ranging from 13 to 23 years of age. The current study endeavors to build upon the knowledge base in this area by offering DBT to youth with and/or at familial risk for BD at CAMH with an emphasis on predictors and mediators of treatment outcomes, with the eventual goal of personalizing treatment selection and delivery. While DBT bodes favorably as a treatment for youth with BD, the literature in this area remains sparse. Moreover, the investigators do not yet understand what clinical characteristics and pre-treatment variables predict and mediate treatment outcomes. There is substantial between-person and within-person variability among youth with and/or at familial risk for BD in terms of risk indicators, type and severity of symptoms, associated distress, and compounding functional impairment. The current study proposes to move beyond questions of efficacy toward identifying individual characteristics that are differentially associated with response to DBT. Identification of baseline demographic and clinical characteristics that are associated with response to DBT (i.e., predictors), as well as time-varying characteristics during the course of treatment (i.e., mediators), could guide iterative optimization of DBT through individualized modifications. Patient engagement will be sought through consultation forums after they have completed the study. Overall, this research endeavors to begin to examine the patient factors that predict and mediate an individual's response to DBT, with important questions to consider, such as: For which youth with and/or at familial risk for BD does this intervention have the greatest effect? Does the intervention have similar effects across sub-groups of youth with BD? The investigators anticipate that the identification of predictor and mediating variables has the potential to inform the iterative personalization of DBT for youth with and/or at familial risk for BD in the future, including content, timing, and relative emphasis on various aspects of DBT (e.g., psychoeducation, skills, individual sessions, family involvement, phone coaching).

ELIGIBILITY:
Inclusion Criteria:

1) English-speaking; 2) Age 13 years, 0 months to 23 years, 11 months; 3) Meet diagnostic criteria for BD by KSADS-PL (< 20 years of age) or SCID-5-RV (> 20 years of age) OR have a biological parent/sibling with BD (type I or II) confirmed via KSADS-PL or SCID-5-RV; 4) If BD-I, taking ≥1 mood stabilizing medication (i.e., antimanic anticonvulsant, antipsychotic, and/or lithium); 5) Followed by a psychiatrist who provides ongoing care; 6a) At least 1 suicide attempt in the past year (actual, interrupted, and/or aborted as measured by the C-SSRS) OR at least 1 preparatory act or behavior in the past year as measured by the C-SSRS OR non-suicidal self-injurious (NSSI) behaviors in the past 3 months (as measured by the C-SSRS) -OR- 6b) Meet youth threshold for at least 2 impulsive behavior categories on question #4 from the SIDP-IV or 1 category is identified as severe (through case discussion that will focus on level of risk, persistence, and impairment); 7) Able and willing to give informed consent/assent to participate.

Exclusion Criteria:

1) Evidence of mental retardation, moderate to severe autism spectrum disorder, or organic central nervous system disorder by the K-SADS-PL (< 20 years of age), parent report, medical history, or school records that would interfere with active participation in DBT; 2) A life-threatening medical condition requiring immediate treatment; 3) Current victim of sexual or physical abuse; 4) Current substance use disorder other than mild cannabis or alcohol use disorder.

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | Baseline to 6 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | 6 months to 12 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | Baseline to 3 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 3 months to 6 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 6 months to 9 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 9 months to 12 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | Baseline to 3 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 3 months to 6 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 6 months to 9 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 9 months to 12 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | Baseline to 6 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | 6 months to 12 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline to 6 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 6 months to 12 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | Baseline to 3 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 3 months to 6 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 6 months to 9 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 9 months to 12 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Treatment Satisfaction Questionnaire (18-item) | 3 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 6 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 9 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 12 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Change in affective lability using the Children's Affective Lability Scale (CALS) | Baseline to 3 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 3 months to 6 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 6 months to 9 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 9 months to 12 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | Baseline to 3 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 3 months to 6 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 6 months to 9 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 9 months to 12 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in functioning using the Children's Global Assessment Scale (C-GAS) or Global Assessment of Functioning (GAF) | Baseline to 6 months
  The Children's Global Assessment Scale (C-GAS) is an adaptation of the Global Assessment of Functioning Scale (GAF) developed to reflect the lowest level of functioning for a child or adolescent during a specified time period. Scores can range from 1-100, with scores above 70 designated as indicating normal functioning. This scale was found to be reliable between interviewers across time. Also, it has demonstrated both discriminant and concurrent validity. This will be completed for participants aged 19 and younger.
  The GAF is a scale originally included in the Diagnostic and Statistical Manual of Mental Disorders (DSM; 4th edition), and is used to rate adult participants' lowest and highest level of functioning in the past year, as well as their current level. It has been found to be reliable and valid. This will be completed for participants aged 20 and older.
Change in functioning using the Children's Global Assessment Scale (C-GAS) or Global Assessment of Functioning (GAF) | 6 months to 12 months
  The Children's Global Assessment Scale (C-GAS) is an adaptation of the Global Assessment of Functioning Scale (GAF) developed to reflect the lowest level of functioning for a child or adolescent during a specified time period. Scores can range from 1-100, with scores above 70 designated as indicating normal functioning. This scale was found to be reliable between interviewers across time. Also, it has demonstrated both discriminant and concurrent validity. This will be completed for participants aged 19 and younger.
  The GAF is a scale originally included in the Diagnostic and Statistical Manual of Mental Disorders (DSM; 4th edition), and is used to rate adult participants' lowest and highest level of functioning in the past year, as well as their current level. It has been found to be reliable and valid. This will be completed for participants aged 20 and older.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | Baseline to 3 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 3 months to 6 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 6 months to 9 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 9 months to 12 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in family functioning using the Family Adaptability and Cohesion Evaluation Scale, IV (FACES-IV) | Baseline to 3 months
  The Family Adaptability and Cohesion Evaluation Scale (FACES-IV) was developed to evaluate the adaptability and cohesion dimensions in family interactions. Youth and parents will complete this self-report questionnaire. Six scales were developed, with two balanced scales and four unbalanced scales designed to tap low and high cohesion (disengaged and enmeshed) and flexibility (rigid and chaotic). Ratio scores above 1 indicate healthier families whereas ratio scores below 1 indicate more problematic families. The six scales in FACES-IV were found to be reliable and valid. Additionally, high levels of concurrent, construct, and discriminant validity were found.
Change in family functioning using the Family Adaptability and Cohesion Evaluation Scale, IV (FACES-IV) | 3 months to 6 months
  The Family Adaptability and Cohesion Evaluation Scale (FACES-IV) was developed to evaluate the adaptability and cohesion dimensions in family interactions. Youth and parents will complete this self-report questionnaire. Six scales were developed, with two balanced scales and four unbalanced scales designed to tap low and high cohesion (disengaged and enmeshed) and flexibility (rigid and chaotic). Ratio scores above 1 indicate healthier families whereas ratio scores below 1 indicate more problematic families. The six scales in FACES-IV were found to be reliable and valid. Additionally, high levels of concurrent, construct, and discriminant validity were found.
Change in family functioning using the Family Adaptability and Cohesion Evaluation Scale, IV (FACES-IV) | 6 months to 9 months
  The Family Adaptability and Cohesion Evaluation Scale (FACES-IV) was developed to evaluate the adaptability and cohesion dimensions in family interactions. Youth and parents will complete this self-report questionnaire. Six scales were developed, with two balanced scales and four unbalanced scales designed to tap low and high cohesion (disengaged and enmeshed) and flexibility (rigid and chaotic). Ratio scores above 1 indicate healthier families whereas ratio scores below 1 indicate more problematic families. The six scales in FACES-IV were found to be reliable and valid. Additionally, high levels of concurrent, construct, and discriminant validity were found.
Change in family functioning using the Family Adaptability and Cohesion Evaluation Scale, IV (FACES-IV) | 9 months to 12 months
  The Family Adaptability and Cohesion Evaluation Scale (FACES-IV) was developed to evaluate the adaptability and cohesion dimensions in family interactions. Youth and parents will complete this self-report questionnaire. Six scales were developed, with two balanced scales and four unbalanced scales designed to tap low and high cohesion (disengaged and enmeshed) and flexibility (rigid and chaotic). Ratio scores above 1 indicate healthier families whereas ratio scores below 1 indicate more problematic families. The six scales in FACES-IV were found to be reliable and valid. Additionally, high levels of concurrent, construct, and discriminant validity were found.
Number, frequency, and type of therapy sessions | At the end of study completion (five years)
  The Therapy Tracking Form will be used to document the date of the therapy session, type of session, session duration, content, and scheduled date for next therapy visit. This form will be completed by the study therapist after each therapy session.

SECONDARY OUTCOMES:
Childhood Trust Events Survey (CTES) | Baseline
  Youth will complete the Childhood Trust Events Survey (CTES) long-form, adolescent version, a 30-item self-report screening survey that assesses exposure to adversity across a breadth of domains including physical, emotional, and sexual abuse; alcohol/drug users in home; family members in prison; caregiver with mental illness; domestic violence; loss/separation from caregiver; and other traumatic events. In addition, the CTES queries the age and perceived intensity of each type of adversity. Parents will complete the caregiver version of the CTES, a 26-item survey that asks if their child has been exposed to the same domains of adversity as queried in the adolescent version.
Change in parental psychological distress using the Symptom Checklist-90 (SCL-90) | Baseline to 3 months
  The Symptom Checklist-90 (SCL-90) is 90-item parent-reported measure used to assess symptoms and complaints that parents may have. It assesses the following dimensions: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and other.
Change in parental psychological distress using the Symptom Checklist-90 (SCL-90) | 3 months to 6 months
  The Symptom Checklist-90 (SCL-90) is 90-item parent-reported measure used to assess symptoms and complaints that parents may have. It assesses the following dimensions: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and other.
Change in parental psychological distress using the Symptom Checklist-90 (SCL-90) | 6 months to 9 months
  The Symptom Checklist-90 (SCL-90) is 90-item parent-reported measure used to assess symptoms and complaints that parents may have. It assesses the following dimensions: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and other.
Change in parental psychological distress using the Symptom Checklist-90 (SCL-90) | 9 months to 12 months
  The Symptom Checklist-90 (SCL-90) is 90-item parent-reported measure used to assess symptoms and complaints that parents may have. It assesses the following dimensions: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and other.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada